CLINICAL TRIAL: NCT06303609
Title: Effects of Non-ablative Radiofrequency on Female Genito-pelvic Pain Disorder: Randomized Clinical Trial
Brief Title: Effects of Non-ablative Radiofrequency on Female Genito-pelvic Pain Disorder
Acronym: Pelvic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Atenção ao Assoalho Pélvico (Other)
Responsible Party: Principal Investigator, Patricia Lordelo, Head of the CentroAAP, Centro de Atenção ao Assoalho Pélvico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 61102222.5.0000.5544
Record Dates: First submitted 2023-11-28; First posted 2024-03-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Pain
Keywords: genito-pelvic pain disorder; radiofrequency; nonablative radiofrequency; women
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency group (Experimental): Once a week, for 8 weeks, patient will undergo monopolar non-ablative radiofrequency application by a trained researcher.
  Interventions: Device: nonablative radiofrequency; Device: Vaginal dilator
- Sham group (Active Comparator): Once a week, for 8 weeks, patient will undergo monopolar non-ablative radiofrequency application by a trained researcher, but the radiofrequency device will not emit the radiofrequency wave.
  Interventions: Device: Vaginal dilator; Device: Sham nonablative radiofrequency

INTERVENTIONS:
Device: nonablative radiofrequency — The active electrode from the nonablative radiofrequency will be applied to the urogenital- and uroanal trigone and the dispersive electrode will be attached to the back of the patient. The water-soluble gel will be applied to the active electrode and to the non-lubricated condom which will involve the electrode. There will be a gradual increase in temperature, monitored by a digital infrared thermometer, to reach temperature between 36°C and 38°C, keeping the movement for two minutes in each area, spending in total around 10 minutes.
  Arms: Radiofrequency group
Device: Vaginal dilator — Both groups will use the vaginal dilator at the end of each session for 15 minutes and all patients will be advised to use it for 15 minutes daily in a home based treatment.
Device: Sham nonablative radiofrequency — The active electrode from the nonablative radiofrequency will be applied to the urogenital- and uroanal trigone and the dispersive electrode will be attached to the back of the patient. The water-soluble gel will be applied to the active electrode and to the non-lubricated condom which will involve the active electrode. As the device will not deliver the radiofrequency wave, the gel will be heated so the patient has the feeling of the temperature change, keeping the movement for two minutes in each area, spending in total around 10 minutes.
  Arms: Sham group

SUMMARY:
The goal of this randomized clinical trial is to verify the response of genito-pelvic pain disorders in women associated with inability to penetrate to the treatment with non-ablative radiofrequency. The main question it aims to answer is: Does non-ablative radiofrequency have a positive effect on the symptoms of genito-pelvic pain disorders associated with inability to penetrate? Before starting the intervention and at one week, one-, three- and six months after the end of the study, participants will be evaluated with 03 questionnaires (Female Sexual Function Index, Sexual Quality of Life and Perceived Stress Scale-10) and will score the visual analogue scale the level of pain with the penetration (from 0 to 10); participants will then undergo digital evaluation of the pelvic floor muscles, using vaginal dilators and electromyographic evaluation. After being randomized, participants will be divided into the Experimental Group and the Sham Group, being submitted to • the use of non-ablative radiofrequency in the anal and urogenital triangles, • the positioning of the vaginal dilator at the end of each session • and participants will be instructed to use the vaginal dilator at home daily. The researchers will compare the groups in relation to the ability to penetrate with reduced vaginal pain, sexual function, quality of sexual life and the correlation between pelvic muscle activity and perceived stress.

DETAILED DESCRIPTION:
Initially, all women included in the study will be briefly and clearly instructed about genito-pelvic pain dysfunction and the anatomy of the pelvic floor. Then the participants will respond to the questionnaires FSFI (Female Sexual Function Index), SQoL-F (Scale of Female Sexual Quality of Life) and the PSS-10 (Perceived Stress Scale - 10).

The FSFI assesses the female sexual function index in the following domains: desire, arousal, lubrication, orgasm, satisfaction and pain. It is self-administered, contains 19 items, with an average response time of nine minutes and addresses aspects of the last four weeks. It is a measure to be considered a potential "gold standard" for evaluating therapeutically induced changes in female sexual function.

The SQoL-F measures the impact of female sexual dysfunctions on women's quality of life, addressing the items: psychosexual feelings, sexual and relationship satisfaction, self-invalidation and sexual repression. It is self-administered, contains 18 items, with an average response time of seven minutes and addresses aspects of the last four weeks.

The EPS-10 measures the degree of stress perceived by individuals within 30 days. It is validated in several countries in versions with 14 questions, 10 questions and four questions. The version with 10 questions was chosen for this study and is self-administered. The scale checks how much respondents evaluate their lives in terms of unpredictability, overload and lack of control, factors recognized as the most relevant factors in cases of stress.

After completing this first process, an Admission Form will be completed in two consecutive stages. In the first stage, the participant will be taken to a reserved location accompanied by at least one properly trained researcher, where questions 1 to 23 of the Admission Form will be answered, in which the following will be collected: demographic data, data social conditions, comorbidities, history of current and previous illness, gynecological history, obstetric history and fecal history, with application of the Rome III Criteria, Bristol Scale, and Visual Analogue Scale (VAS) related to pain during vaginal penetration.

Once the first stage of the Admission Form has been completed, the second stage will begin, in which the participant will be taken to a private office, where will be positioned in the supine position on a stretcher, with the pelvic region uncovered, the lower limbs abducted and flexed for perineal assessment. A trained researcher will carry out the physical evaluation through pelvic inspection and digital vaginal palpation, following the ICS recommendations, for using the letters P, E, R and F of the PERFECT Scheme, associated with a subjective assessment of coordination, use of accessory muscles and symmetry. The findings will be recorded in items 24 to 29 of the Admission Form.

Pelvic floor (PF) EMG will be performed using self-adhesive surface electrodes (Hydrogel Adhesive Electrode 4.5 x 3.8cm, Meditrace 200, Kendal™, Mansfield - USA) connected to an Electromyography (EMG) device (New Miotool Uro™, Miotec, Porto Alegre - BR) which converts the myoelectric signal into values expressed in microvolts (μV). EMG data will be collected and analyzed using Miotec Suite version 1.0 software (Miotec®, Porto Alegre, Brazil). In this software, the 20Hz high-pass, 500Hz low-pass and 60Hz notch filters will be used and the data can be viewed in the form of graphs. To perform the technique, the following materials will be needed: five surface electrodes, adhesive tape, 70% alcohol, paper towel and 2 pairs of gloves. 02 (two) surface electrodes will be attached, in the perianal region (positioning equivalent to 2 and 8 on the clock), 02 (two) on the trunk of the right external oblique muscle (to evaluate the abdominal muscles) and 01 (one) on the diaphysis of the right clavicle. To place the electrode in the perianal region, the patient is positioned in lateral decubitus with the lower limbs adducted and flexed. To place the electrode on the right external oblique muscle, the patient is positioned in DD with lower limbs extended and this muscle is asked to contract with trunk flexion and rotation to the left.

The examination will be carried out in two moments: the first moment with the patient in the supine position (DD) and in the second moment, in orthostasis. Initially, in DD, with the lower limbs extended, the EMG assessment will capture the Maximum Voluntary Contraction (MVC). 03 maximum contractions of the PFM (pelvic floor muscles) will be requested and the average of the 03 (three) contractions will be recorded. After recording the MVC, the collection of PF muscle activity in DD begins.

Collection 01: Starts with the collection of basal electrical activity for 30 seconds. The verbal command will be: "Keep your anus relaxed." The participant will then be asked to perform five tonic contractions (CT). The volunteer will be instructed to perform five contractions maintained for 10 seconds and the same relaxation time. The evaluator will determine when to contract and relax. The verbal command will be: "Contract your anus as if you were holding back a fart and hold for 10 seconds and then relax for the same amount of time. Do this five times following my voice command (Contract, hold, hold, hold... and relax.)." When finished, the participant will have to rest for 30 seconds. Finally, you will be asked to perform 10 maximum contractions of 1 second with complete relaxation between them (phasic contractions). The verbal command will be: "Contract your anus as if you were holding back a fart and relax. Do this ten times following my voice command (Contract, relax, contract, relax...)". After the phasic contractions, ask the patient to rest for ten seconds to complete the collection.

Collection 02: All the steps of collection 01 are repeated, but the orthostasis position will be adopted with the upper limbs along the body. All EMG collection will be recorded and analyzed by the Miotec Suite software version 1.0 (Miotec®, Porto Alegre, Brazil) and stored on a portable computer. During the entire examination, dynamic inspection will also be carried out (visual and by EMG, simultaneously) evaluating the presence of visible contraction of the PF muscles, the presence of contraction of other muscles (gluteus maximus, thigh adductors and abdominal muscles) and the visible relaxation capacity (good, regular, incomplete or absent).

After initial assessment, all patients will be randomized, using a random table generated in the program available on the website: www.random.org into two groups: a Radiofrequency Group (RG) made up of 28 women and a Control Group (CG) made up of by 28 participants. The volunteers who will be part of the GR group will receive physiotherapeutic treatment through the application of non-ablative RF with the aim of promoting perineal muscle relaxation. In each session, which will take place once a week, the patient will be taken to a private office and will be positioned in the supine position on a stretcher, with the pelvic region uncovered, the lower limbs abducted and flexed for the application of non-ablative RF through a trained researcher.

In women in the CG group, the device for applying non-ablative RF will be turned off and the conduction gel will be heated by a resistor. The remainder of the protocol will be identical to that of the RG group. Only the researcher who performed the procedure will know which group the patient belongs to, with allocation confidentiality being maintained for the other researchers and for the patient. Immediately after the application of RF, both in the RG group and in the CG group, a researcher who will not know which group the patient belongs to will try to introduce a lubricated vaginal dilator for 15 minutes, with the aim of promoting stretching of vaginal introitus.

There are six sizes of vaginal dilator that will be changed gradually with each session, depending on the patient's acceptability. In this study, the ABSOLOO vaginal dilator set will be used, which contains six devices with different colors and sizes: green nº 1: diameter 1.16cm, length 6.5cm; rose nº 2: diameter 1.90cm, length 7.5cm; yellow nº 3: diameter 2.15cm, length 8.7cm; purple nº 4: diameter 2.5cm, length 10.9cm; blue nº 5: diameter 3.10cm, length 13.20cm; and orange nº 6: diameter 3.5cm, length 14.5cm. The last size of vaginal dilator will be the one chosen by the patient. After the procedure, the patient will be instructed to exercise with the dilator at home daily for 15 minutes.

At the end of each session, the following will be recorded in the Monitoring Sheet: the tolerance of digital vaginal insertion, the size of the current dilator, the perception of VAS related to pain during vaginal penetration and the LIKERT scale of satisfaction in relation to the RF treatment . Eight RF application sessions will be held, weekly, totaling a period of two months.

One week after the last session, the final reassessment will be carried out, in which the participant will be taken to a private office, will be positioned in the supine position on a stretcher, with the pelvic region uncovered, the lower limbs abducted and flexed for the perineal assessment. and a trained researcher will carry out the evaluation through inspection, vaginal digital palpation, following the ICS recommendations, to use the letters P, E, R and F of the PERFECT Scheme associated with an evaluation as well. subjective coordination, use of accessory muscles and symmetry. An ABSOLOO vaginal dilator of the size chosen by the patient will be inserted and an electromyographic evaluation will be carried out.

The findings will be recorded in the Reassessment Form: tolerance of digital vaginal insertion, the size of the current dilator, the perception of VAS related to pain during vaginal penetration and the LIKERT scale of satisfaction in relation to treatment with RF. The FSFI, SQoL-F and EPS-10 instruments will also be answered again. After treatment, a follow-up period of one, three and six months will be carried out, when the Reassessment Form and the FSFI, SQoL-F and EPS-10 instruments will be reapplied.

If the patient does not attend the reevaluations, telephone contact will be made and the FSFI, SQoL-F and EPS-10 will be applied remotely. RF treatment will be considered successful based on the patient's ability to have sexual intercourse including complete penetration of the penis followed by the partner's ejaculation, without complaining of pain.

ELIGIBILITY:
Inclusion Criteria:

* Women with genito-pelvic pain disorder associated to penetration.

Exclusion Criteria:

* Chronic degenerative disease
* Cognitive impairment
* Genital agenesis
* History of vaginal cancer or genital radiotherapy
* Pelvic or lumbosacral prostheses
* Cardiac pacemakers
* Pregnant women
* Infections in the genital or systemic region
* Any type of treatment for genito-pelvic pain disorder
* Unstable relationship with the same partner
* Partner with sexual complaints.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-04-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Penetration capacity with reduced vaginal pain | From enrollment till 6 months after the end of treatment: at the assessment, before each session (8 sessions, one per week), one week after the last session, one, three and six months after the end of the treatment
  To assess the primary outcome it will be used the Visual Analogue Scale (VAS) related to pain during vaginal penile penetration and during the vaginal dilatator penetration. The score varies from 0 (no pain) to 10 (maximum pain). Diminishing at least 2 points on the scale means positive diffence with the treatment. Also the change of the size of the vaginal dilatator will be a measure to positive response to the treatment. There are 6 sizes: green nº 1: diameter 1.16cm, length 6.5cm; rose nº 2: diameter 1.90cm, length 7.5cm; yellow nº 3: diameter 2.15cm, length 8.7cm; purple nº 4: diameter 2.5cm, length 10.9cm; blue nº 5: diameter 3.10cm, length 13.20cm; and orange nº 6: diameter 3.5cm, length 14.5cm

SECONDARY OUTCOMES:
Sexual function | From enrollment till 6 months after the end of treatment: at the assessment, before each session (8 sessions, one per week), one week after the last session, one, three and six months after the end of the treatment
  To measure the change in the sexual function it will be use the Female Sexual Function Index. It consists of 19 items and the score varies from 2 to 36. A score below or equal to 26 indicates sexual dysfunction.
Quality of sexual life | From enrollment till 6 months after the end of treatment: at the assessment, before each session (8 sessions, one per week), one week after the last session, one, three and six months after the end of the treatment
  To measure the change in quality of sexual life it will be used the Scale of Female Sexual Quality of Life. It consists of 18 items, rated using a six-point scale (completely agree to completely disagree). The total score can range from 18 to 108 points. Higher scores indicate better female sexual quality of life.
Stress perception | From enrollment till 6 months after the end of treatment: at the assessment, before each session (8 sessions, one per week), one week after the last session, one, three and six months after the end of the treatment
  To measure the stress perception it will be used the Stress Perception Scale - 10. There are 10 items and the total score can range from 0 to 40. The higher scores indicate higher levels of perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Atenção ao Assoalho Pelvico, Salvador, Estado de Bahia, Brazil